CLINICAL TRIAL: NCT07107906
Title: The CONNECT Program: Engaging Community Organizations in the Implementation and Evaluation of a Group Telehealth Mental Health Program for Older Canadians
Brief Title: Evaluating and Implementing The CONNECT Program - a Group-Based Telehealth Intervention to Reduce Social Isolation, Loneliness, and Mental Health Symptoms in Adults Ages 55+, Compared to Routine Community-Based Programming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: A & O: Support Services for Older Adults (Unknown); Brella Community Services Society (Unknown); Senior Citizens Assistance Program (Unknown); CHI - Centre for Healthcare Innovation (Unknown)
Responsible Party: Principal Investigator, Kristin Reynolds, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HE2024-0150; 58465 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Loneliness; Social Isolation; Depression Disorders; Anxiety
Keywords: Psychological Flexibility; Loneliness; Social Isolation; Anxiety; Depression; Older adult; Aged; Psychotherapy, Group; Acceptance and Commitment Therapy; Mental Health; Telemedicine; Mental Health Teletherapy; Community Mental Health Services; Community-Based Participatory Research; Program Evaluation; Randomized Controlled Trial; Implementation Effectiveness Hybrid Design; Cross-Over Studies
MeSH Terms: conditions — Social Isolation; Anxiety Disorders; Depression; Psychological Well-Being | interventions — Community Participation

STUDY DESIGN:
Intervention Model Description: Participants within each community site will be randomized to one of two sequences: (1) The CONNECT Program followed by community programming as usual, or (2) community programming as usual followed by The CONNECT Program. Each phase consists of a 6-week intervention. After the first phase, participants will cross over to receive the alternative condition. All participants will receive both interventions during the study period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A non-affiliated researcher will generate the randomization sequence and assign participant IDs to one of two intervention sequences (the CONNECT program - Community programming as usual or Community programming as usual - the CONNECT program) prior to recruitment. Each participant will be assigned a unique ID, and outcome data will be collected and analyzed using only these IDs. The study coordinator will be unblinded to group assignment for the purpose of managing recruitment, scheduling, and follow-up assessments. However, outcome investigator responsible for analyzing primary, secondary and other pre-specified outcomes will remain blinded to group allocation and will use de-identified datasets for analysis. The outcome assessors responsible for collecting baseline, post-intervention, and follow-up data are blinded in this study. Participants, facilitators, and the study coordinator will not be blinded due to the nature of behavioral interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The CONNECT Program first (Experimental): Participants in this arm will receive The CONNECT Program during the first 6-week phase, followed by community participation as usual during the second 6-week phase.
  Interventions: Behavioral: The CONNECT Program; Behavioral: Community Participation as Usual (Service as Usual)
- Community-based programming as usual (Service as Usual) first (Active Comparator): Participants in this arm will receive community participation as usual during the first 6-week phase, followed by The CONNECT Program during the second 6-week phase. Community participation as usual refers to the regular group programs already offered by community organizations in-person, over the phone or virtually.
  Interventions: Behavioral: The CONNECT Program; Behavioral: Community Participation as Usual (Service as Usual)

INTERVENTIONS:
Behavioral: The CONNECT Program — A group-based telehealth intervention grounded in Acceptance and Commitment Therapy (ACT), self-compassion, and successful aging theories, aimed at reducing social isolation, loneliness, and mental health symptoms among adults 55+. Delivered over six weeks via group phone or Zoom sessions. The CONNECT Program includes 6 weekly 90-minute group sessions, with structured workbooks and homework. The CONNECT Program is delivered in two modalities (group telephone or Zoom videoconferencing).
Behavioral: Community Participation as Usual (Service as Usual) — These community-based programs may include social, educational, or recreational group sessions that are already offered by local organizations - either in person, by phone, or virtually.

SUMMARY:
Older adults in Canada are experiencing increasing levels of social isolation, loneliness, and mental health challenges, including anxiety and depression - trends that have worsened during and following the COVID-19 pandemic. Research consistently shows that loneliness and social isolation are associated with poorer mental and physical health outcomes, increased risk of dementia, and increased mortality. At the same time, social connection has a strong protective impact on health and well-being. Community-based programs that promote both social engagement and psychological support are urgently needed, particularly since older adults are less likely to access formal mental health services.

Approximately 3-11% of older adults meet diagnostic criteria for mood or anxiety disorders each year, with even more experiencing elevated symptoms that greatly influence quality of life. Subsyndromal depression in late life is estimated to occur two to three times more often than major depressive disorder. Despite these needs, up to 70% of older adults with anxiety or mood disorders do not access psychological services, often due to low mental health literacy or practical barriers to care. At the same time, participation in community activities is associated with improved emotional well-being, greater social support, and lower rates of depression and anxiety.

To bridge this need for support, our team developed and pilot-tested The CONNECT Program - a group-based mental health intervention for adults 55 years and older, delivered via telephone or virtually. The CONNECT Program is grounded in Acceptance and Commitment Therapy (ACT), self-compassion, and theories of successful aging, and aims to improve psychological flexibility; reduce loneliness, social isolation, and co-occurring symptoms of depression and anxiety. A Manitoba pilot study (N = 34) demonstrated promising outcomes in terms of feasibility, acceptability, and preliminary effectiveness with the telephone-based group intervention.

The current trial will evaluate the implementation and effectiveness of The CONNECT Program in four Canadian provinces (British Columbia, Manitoba, New Brunswick, Saskatchewan), using an implementation-effectiveness hybrid design and a crossover randomized controlled trial. This study compares The CONNECT Program, delivered via telephone or virtually, to routine community programming (i.e., community participation as usual), which may occur in telephone, virtual, or in-person formats. The primary outcome is psychological flexibility; secondary outcomes include loneliness, social isolation, anxiety, depression, emotional support, mental health literacy. Implementation outcomes will be evaluated following the Proctor et al. framework.

This trial will contribute evidence on the mental health needs of adults 55+ and the value of low-barrier, community-based programs delivered remotely. Findings will guide further national and international implementation of The CONNECT Program and similar initiatives aimed at addressing the challenges of loneliness, social isolation, and mental health problems in late life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 years or older
* Able to speak, read, and understand English
* Can manage hearing or vision changes well enough to participate in group conversations
* Self-reported experiences of loneliness, social isolation, and/or mental health challenges (e.g., anxiety or depressive symptoms)

Exclusion Criteria:

* Cannot communicate in English (verbal or written)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Flexibility from Baseline (Acceptance and Action Questionnaire-II) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Psychological flexibility will be measured using the Acceptance and Action Questionnaire-II, a 7-item self-report scale. Scores range from 7 to 49, with higher scores indicating greater psychological inflexibility, and lower scores indicating greater psychological flexibility. Psychological flexibility is a core target of Acceptance and Commitment Therapy and has been shown to be a transdiagnostic mechanism of change in psychotherapy outcomes.

SECONDARY OUTCOMES:
Change in Loneliness from Baseline (DeJong Gierveld Loneliness Scale) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Loneliness will be assessed using the De Jong Gierveld Loneliness Scale, a validated 6-item self-report instrument designed to measure emotional and social dimensions of loneliness. Total scores range from 0 to 6, with higher scores indicating greater loneliness and lower scores indicating less loneliness. Loneliness is a key risk factor for late-life depression and anxiety and is associated with negative physical and cognitive health outcomes.
Change in Social Isolation from Baseline (PROMIS Social Isolation 8a) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Social isolation will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation 8a short form, an 8-item standardized measure of perceived disconnection from others. Scores range from 8 to 40, with higher scores indicating greater social isolation. Social isolation is an objective risk factor for poor mental and physical health and is closely linked to late-life depression, anxiety, and cognitive decline.
Change in Emotional Support from Baseline (PROMIS Emotional Support) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Emotional support will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support Short Form, a standardized self-report measure evaluating the perceived availability of caring and understanding individuals in one's life. Scores range from 4 to 20, with higher scores indicating greater emotional support. Greater emotional support is associated with reduced risk of depression, better coping with stress, and improved quality of life in older adults.
Change in Anxiety Symptoms from Baseline (PROMIS Anxiety Short Form 4a) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Anxiety symptoms will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 4a, a validated 4-item self-report scale capturing core features of anxiety such as fear, worry, and nervousness. Scores range from 4 to 20, with higher scores indicating greater severity of anxiety symptoms. Anxiety is prevalent among older adults and is strongly linked to social isolation and reduced quality of life.
Change in Depressive Symptoms from Baseline (PROMIS Depression Short Form 4a) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Depressive symptoms will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 4a, a 4-item self-report measure capturing core features such as sadness, hopelessness, and lack of interest in activities. Scores range from 4 to 20, with higher scores indicating greater severity of depressive symptoms. Subsyndromal depressive symptoms are common in late life and are associated with lower quality of life and increased health risk.
Change in Mental Health Literacy from Baseline (Brief Mental Health Literacy Scale) | At baseline (Week 0), after community-based programming as usual if delivered first (Week 6), after the CONNECT program (Week 6 or 12 depending on sequence), and at 6-month follow-up (Week 30-36).
  Mental health literacy will be assessed using the Brief Mental Health Literacy Scale. This 4-item self-report measure evaluates perceived knowledge about signs and symptoms, possible causes, types of professional help available, and how to seek help for common mental health problems (e.g., anxiety, depression). Respondents rate their knowledge on a 5-point Likert scale (1=not at all, to 5=extremely). Composite scores range from 4 to 20, with higher scores indicating greater perceived mental health literacy. Older adults typically have lower mental health literacy than younger groups, which may hinder service use and self-identification of mental health problems.

OTHER OUTCOMES:
Acceptability of the CONNECT Program: Post-Program Survey | Once post-program (at Week 6 or Week 12, depending on intervention sequence).
  Acceptability is defined as the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Acceptability of the CONNECT Program will be assessed using a post-program survey that includes both Likert-scale items (1=not at all acceptable to 5=completely acceptable, with higher scores indicating greater acceptability) and open-ended questions. Survey items were developed based on the Proctor implementation outcomes framework.
Acceptability of the CONNECT Program: Intervention Content Evaluation | Once post-program (Week 6 or Week 12).
  Participant ratings of the CONNECT program intervention content acceptability will be assessed using the Intervention Content Evaluation survey adapted from McCracken et al., 2014. This survey includes Likert ratings of key aspects of the intervention. Items are rated on a 3-point scale: satisfied, neither satisfied nor not satisfied, or not satisfied. Higher satisfaction across items reflects greater acceptability of the CONNECT program content.
Acceptability of the CONNECT Program: Exit Interview | Once post-program (at Week 6 or Week 12).
  Qualitative exit interviews assessing participants' perceptions and overall satisfaction with the CONNECT Program. Data will be analyzed thematically to identify patterns in participant experience.
Acceptability of the CONNECT Program: Group Session Rating Scale | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Weekly participant ratings of the quality and acceptability of group sessions will be assessed using the Group Session Rating Scale. This brief self-report measure captures participants' perceptions of four key aspects of each session: relationship, goals and topics, approach or method, and overall experience. Each item is rated on a 10-point visual analog scale, with higher scores indicating greater session acceptability.
Acceptability of the CONNECT Program: Intervention Delivery Type Evaluation | Once post-program (Week 6 or Week 12).
  Participant ratings of CONNECT program intervention delivery mode satisfaction and usability will be assessed using the Intervention Delivery Type Evaluation adapted from McCracken et al., 2014. Responses are provided using a 3-point Likert scale: satisfied, neither satisfied nor not satisfied, and not satisfied. Higher ratings reflect greater delivery acceptability; lower ratings reflect challenges or dissatisfaction with the delivery mode.
Acceptability of the CONNECT Program: Weekly Facilitator Check-in Questionnaire | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Acceptability will be evaluated through weekly facilitator-reported tracking of acceptability indicators such as attendance, dropout rates, reasons for missing sessions or discontinuing participation using the weekly facilitator check-in questionnaire (developed for this trial).
Adoption of the CONNECT Program: Post-Program Survey | Once post-program (Week 6 or Week 12, depending on intervention sequence).
  Adoption is defined as the intention, initial decision, or action to employ or continue using the CONNECT Program. Adoption will be assessed using a post-program survey, each item rated on a 5-point Likert scale (1=Not at all 5=Extremely), and open-ended questions (items developed based on Proctor implementation framework).
Adoption of the CONNECT Program: Weekly Facilitator Check-in Questionnaire | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Adoption will be evaluated through weekly facilitator-reported tracking of adoption indicators such as attendance, dropout rates, reasons for missing sessions or discontinuing participation using the weekly facilitator check-in questionnaire (developed for this trial).
Appropriateness of the CONNECT Program: Post-Program Survey | Once post-program (Week 6 or Week 12, depending on intervention sequence).
  Appropriateness is the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given setting, provider, or consumer, and/or the perceived fit of the innovation to address a particular issue or problem. Data will be collected through the post-program survey item, rated on a 5-point Likert scale (1=Not at all a good fit to 5=Excellent fit). Higher scores reflect greater perceived appropriateness. Participants will also respond to the open-ended question.
Appropriateness of the CONNECT Program: Exit Interview | Once post-program (Week 6 or Week 12).
  Qualitative assessment of participants' perceptions of the CONNECT Program's appropriateness using open-ended interview questions. Data will be analyzed thematically to identify patterns in participant experience.
Appropriateness of the CONNECT Program: Intervention Content Evaluation | Once post-program (Week 6 or Week 12).
  Participants' evaluation of intervention content appropriateness using the Intervention Content Evaluation adapted from McCracken et al. (2014). Participants will rate satisfaction with specific components of the CONNECT Program using a 3-point scale (satisfied, neither satisfied nor not satisfied, not satisfied). Higher ratings across items indicate greater perceived appropriateness of the intervention content; lower ratings reflect poorer perceived fit or relevance.
Appropriateness of the CONNECT Program: Intervention Delivery Type Evaluation | Once post-program (Week 6 or Week 12).
  Participants' perceptions of the appropriateness of the CONNECT Program's delivery mode will be assessed using the Intervention Delivery Type Evaluation Survey, adapted from McCracken et al. (2014). The survey includes participant ratings of specific delivery-related aspects using a 3-point scale (satisfied, neither satisfied nor not satisfied, not satisfied). Higher ratings indicate greater perceived appropriateness and fit of the delivery format.
Appropriateness of the CONNECT Program: Weekly Facilitator Check-in Questionnaire | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Appropriateness will be evaluated through weekly facilitator-reported tracking of appropriateness indicators such as attendance, dropout rates, reasons for missing sessions or discontinuing participation using the weekly facilitator check-in questionnaire (developed for this trial).
Feasibility of the CONNECT Program: Post-Program Survey | Once post-program (Week 6 or Week 12, depending on intervention sequence).
  Feasibility is defined as the extent to which an innovation can be successfully used or carried out within a given agency or setting. Feasibility will be assessed using the post-program survey item, rated on a 5-point Likert scale (1=Not at all manageable to 5=Very manageable). Higher scores indicate greater perceived feasibility. Participants will also respond to the open-ended question.
Feasibility of the CONNECT Program: Exit Interview | Once post-program (Week 6 or Week 12).
  Qualitative assessment of participants' perceptions of the CONNECT Program's feasibility using open-ended interview questions. Data will be analyzed thematically to identify patterns in participant experience.
Feasibility of the CONNECT Program: Intervention Content Evaluation | Once post-program (Week 6 or Week 12).
  Participants' evaluation of intervention content feasibility using the Intervention Content Evaluation adapted from McCracken et al. (2014). Participants will rate satisfaction with specific components of the CONNECT Program using a 3-point scale (satisfied, neither satisfied nor not satisfied, not satisfied). Higher ratings across items indicate greater perceived feasibility of the intervention content; lower ratings reflect poorer perceived feasilibity.
Feasibility of the CONNECT Program: Intervention Delivery Type Evaluation | Once post-program (Week 6 or Week 12).
  Participants' perceptions of the feasibility of the CONNECT Program's delivery mode will be assessed using the Intervention Delivery Type Evaluation Survey, adapted from McCracken et al. (2014). The survey includes participant ratings of specific delivery-related aspects using a 3-point scale (satisfied, neither satisfied nor not satisfied, not satisfied). Higher ratings indicate greater perceived feasibility of the delivery format.
Feasibility of the CONNECT Program: Weekly Facilitator Check-in Questionnaire | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Feasibility will be evaluated through weekly facilitator-reported tracking of feasibility indicators such as attendance, dropout rates, reasons for missing sessions or discontinuing participation using the weekly facilitator check-in questionnaire (developed for this trial).
Penetration of the CONNECT Program | Post-CONNECT program at Week 6 or Week 12, depending on randomization sequence.
  Penetration refers to the integration of an innovation within a service setting and its reach among intended users. At the recipient level, it is defined as the number of eligible individuals who use a service, divided by the total eligible population. At the setting level, it is the number of providers delivering the service, divided by the total number trained or expected to deliver it. Penetration will be assessed using the post-program survey item, rated on a 5-point Likert scale (1=almost none of them to 5=almost all of them). Higher scores indicate greater perceived program reach among eligible individuals. Participants will also respond to an open-ended question.
Implementation Costs of the CONNECT Program | Post-CONNECT program at Week 6 or Week 12, depending on randomization sequence.
  Cost (incremental or implementation cost) is defined as the cost impact of an implementation effort. Implementation cost will be assessed using the post-program survey item, rated on a 5-point Likert scale (1=It was no burden at all to 5=A very big burden). Higher scores indicate greater perceived cost or burden. Participants will also respond to an open-ended question.
Sustainability of the CONNECT Program: Post-Program Survey | Once post-program (Week 6 or Week 12, depending on intervention sequence).
  Sustainability is defined as the extent to which a newly implemented treatment is maintained or institutionalized within a service setting's ongoing, stable operations. Sustainability will be assessed using the post-program survey item, rated on a 5-point Likert scale (1=Not at all sure to 5=Very sure). Higher scores indicate greater perceived sustainability. Participants will also respond to the open-ended question.
Sustainability of the CONNECT Program: Weekly Facilitator Check-in Questionnaire | Weekly during the CONNECT program (Weeks 1-6 or 7-12, depending on sequence).
  Sustainability will be evaluated through weekly facilitator-reported tracking of sustainability indicators such as attendance, dropout rates, reasons for missing sessions or discontinuing participation using the weekly facilitator check-in questionnaire (developed for this trial).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds K, Ceccarelli L, Mackenzie CS. Reliability and validity of a new brief measure of mental health literacy. Presented at: CPA 2020 Virtual Series; 2020.
- [Background] Duncan BL, Miller SD. Group Session Rating Scale. Chicago, IL: International Center for Clinical Excellence; 2007.
- [Background] De Jong Gierveld J, Van Tilburg T. A 6-item scale for overall, emotional, and social loneliness: confirmatory tests on survey data. Res Aging. 2006 Sep;28(5):582-598. doi: 10.1177/0164027506289723.
- [Background] Salinas J, Beiser AS, Samra JK, O'Donnell A, DeCarli CS, Gonzales MM, Aparicio HJ, Seshadri S. Association of Loneliness With 10-Year Dementia Risk and Early Markers of Vulnerability for Neurocognitive Decline. Neurology. 2022 Mar 29;98(13):e1337-e1348. doi: 10.1212/WNL.0000000000200039. Epub 2022 Feb 7. PMID 35131906
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] McCracken LM, Vowles KE, Zhao-O'Brien J. Further development of an instrument to assess psychological flexibility in people with chronic pain. J Behav Med. 2010 Oct;33(5):346-54. doi: 10.1007/s10865-010-9264-x. Epub 2010 May 26. PMID 20502955
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Golden J, Conroy RM, Lawlor BA. Social support network structure in older people: underlying dimensions and association with psychological and physical health. Psychol Health Med. 2009 May;14(3):280-90. doi: 10.1080/13548500902730135. PMID 19444706
- [Background] Harasemiw O, Newall N, Shooshtari S, Mackenzie C, Menec V. From Social Integration to Social Isolation: The Relationship Between Social Network Types and Perceived Availability of Social Support in a National Sample of Older Canadians. Res Aging. 2018 Sep;40(8):715-739. doi: 10.1177/0164027517734587. Epub 2017 Oct 5. PMID 28982271
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Hayes SC, Ciarrochi J, Hofmann SG, Chin F, Sahdra B. Evolving an idionomic approach to processes of change: Towards a unified personalized science of human improvement. Behav Res Ther. 2022 Sep;156:104155. doi: 10.1016/j.brat.2022.104155. Epub 2022 Jul 3. PMID 35863243
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Sibbald B, Roberts C. Understanding controlled trials. Crossover trials. BMJ. 1998 Jun 6;316(7146):1719. doi: 10.1136/bmj.316.7146.1719. No abstract available. PMID 9614025
- [Background] Landes SJ, McBain SA, Curran GM. An introduction to effectiveness-implementation hybrid designs. Psychiatry Res. 2019 Oct;280:112513. doi: 10.1016/j.psychres.2019.112513. Epub 2019 Aug 9. PMID 31434011
- [Background] Reynolds KA, Sommer J, Mackenzie CS, Koven L. A Profile of Social Participation in a Nationally Representative Sample of Canadian Older Adults: Findings from the Canadian Longitudinal Study on Aging. Can J Aging. 2022 Dec;41(4):505-513. doi: 10.1017/S0714980822000150. Epub 2022 Jul 28. PMID 35899988
- [Background] Cohen-Mansfield J, Frank J. Relationship between perceived needs and assessed needs for services in community-dwelling older persons. Gerontologist. 2008 Aug;48(4):505-16. doi: 10.1093/geront/48.4.505. PMID 18728300
- [Background] Berard LDH, Mackenzie CS, Reynolds KA, Thompson G, Koven L, Beatie B. Choice, coercion, and/or muddling through: Older adults' experiences in seeking psychological treatment. Soc Sci Med. 2020 Jun;255:113011. doi: 10.1016/j.socscimed.2020.113011. Epub 2020 Apr 25. PMID 32387873
- [Background] Kessler RC, Merikangas KR, Berglund P, Eaton WW, Koretz DS, Walters EE. Mild disorders should not be eliminated from the DSM-V. Arch Gen Psychiatry. 2003 Nov;60(11):1117-22. doi: 10.1001/archpsyc.60.11.1117. PMID 14609887
- [Background] Meeks TW, Vahia IV, Lavretsky H, Kulkarni G, Jeste DV. A tune in "a minor" can "b major": a review of epidemiology, illness course, and public health implications of subthreshold depression in older adults. J Affect Disord. 2011 Mar;129(1-3):126-42. doi: 10.1016/j.jad.2010.09.015. PMID 20926139
- [Background] Scott T, Mackenzie CS, Chipperfield JG, Sareen J. Mental health service use among Canadian older adults with anxiety disorders and clinically significant anxiety symptoms. Aging Ment Health. 2010 Sep;14(7):790-800. doi: 10.1080/13607861003713273. PMID 20635231
- [Background] Reynolds K, Pietrzak RH, El-Gabalawy R, Mackenzie CS, Sareen J. Prevalence of psychiatric disorders in U.S. older adults: findings from a nationally representative survey. World Psychiatry. 2015 Feb;14(1):74-81. doi: 10.1002/wps.20193. PMID 25655161
- [Background] Byers AL, Arean PA, Yaffe K. Low use of mental health services among older Americans with mood and anxiety disorders. Psychiatr Serv. 2012 Jan;63(1):66-72. doi: 10.1176/appi.ps.201100121. PMID 22227762
- [Background] Mackenzie CS, Reynolds K, Cairney J, Streiner DL, Sareen J. Disorder-specific mental health service use for mood and anxiety disorders: associations with age, sex, and psychiatric comorbidity. Depress Anxiety. 2012 Mar;29(3):234-42. doi: 10.1002/da.20911. Epub 2011 Nov 7. PMID 22065571
- [Background] Cacioppo JT, Hawkley LC, Crawford LE, Ernst JM, Burleson MH, Kowalewski RB, Malarkey WB, Van Cauter E, Berntson GG. Loneliness and health: potential mechanisms. Psychosom Med. 2002 May-Jun;64(3):407-17. doi: 10.1097/00006842-200205000-00005. PMID 12021415
- [Background] Ward M, Briggs R, McGarrigle CA, De Looze C, O'Halloran AM, Kenny RA. The bi-directional association between loneliness and depression among older adults from before to during the COVID-19 pandemic. Int J Geriatr Psychiatry. 2023 Jan;38(1):e5856. doi: 10.1002/gps.5856. PMID 36462183
- [Background] Holt-Lunstad J. A pandemic of social isolation? World Psychiatry. 2021 Feb;20(1):55-56. doi: 10.1002/wps.20839. No abstract available. PMID 33432754
- [Background] Greig F, Perera G, Tsamakis K, Stewart R, Velayudhan L, Mueller C. Loneliness in older adult mental health services during the COVID-19 pandemic and before: Associations with disability, functioning and pharmacotherapy. Int J Geriatr Psychiatry. 2022 Jan;37(1):10.1002/gps.5630. doi: 10.1002/gps.5630. Epub 2021 Oct 6. PMID 34614534
- [Derived] Kudar K, Gopinath G, Ross A, Balshaw R, Chau E, Christianson I, Koven L, Mackenzie CS, Miller S, Newall N, Ouellet L, Sibley K, Sanina A, Wedhorn R, Reynolds KA. Evaluating and implementing The CONNECT Program-A group-based telehealth intervention to reduce social isolation, loneliness, and mental health symptoms in adults 55+ vs routine community programming: Study protocol for a randomized controlled trial. PLoS One. 2025 Nov 11;20(11):e0336031. doi: 10.1371/journal.pone.0336031. eCollection 2025. PMID 41218068